## Evaluation of Preventive (Stay Safe) Training Program of Child Abuse for Teachers and Children: A Randomized Controlled Trial from Multan City

**Protocol of the study** 

By

Zainab Noor Hussain
PSY-07
M.Phil. Applied Psychology

Supervisor

Dr. Rizwana Amin



**Department of Applied Psychology** 

Bahauddin Zakariya University, Multan

Date: September 15, 2018

**Protocol of the study:** 

The protocol of the study covers some steps which describes the phases or session of the

programme undertaking in the study. These are as follows:

Session 1 introducing programme to teachers and children. In the first meeting, informed

consent form is given to children and teachers and introducing the topic briefly. The main

purpose of this session is to inform the participants about their participation in the study and

developing their understanding towards the concept of the topic of research.

Session 2 pre-testing from children and teachers. In the second, demographical data of

children and their parents were collected from children and measure conceptual understanding

of the topics or variables of the study through questionnaire without giving any lessons. This

session basic purpose is to measure the mind set of children and teachers about child abuse

without any discussion to analyze the pre intervention stage of children and teachers. It consist

of pre-testing as scales are applied that measure the level of understanding of children and

teachers about child abuse. Children safety knowledge and skills and self-esteem in regards to

abuse is measured and teacher's attitude and knowledge about abuse is also measured from

teachers. Both control and experimental group pass through this stage called pre-testing.

Session 3 describe programme lessons to children. After collecting pre-testing data from all

participants, as experimental group receives training which consist of Stay Safe Programme

lessons on different topics. In this session, children are being informed about the nature of this

Programme, its context, its content, its tools and tactics and also guide them about their

participation in this Programme. Stay safe Programme consist of 5 to 6 lessons with different

topics that are very sensitive in nature. The topics consist of feelings (feelings of being safe

and unsafe), bullying, touch (appropriate and inappropriate touch), secrets (bad secrets and good secrets) and strangers.

Session 4 stay safe programme lessons for children. In this session, the Stay Safe Programme initiated properly by giving lessons to children about the topic feelings and bullying. By giving different activities to children and show them different pictures about different emotions and feelings of children at different circumstances. It also contain a short story of the girl who face a bad feelings on her birthday party, she faced an incident but she is unable to tell; by telling this story to children encourage them to speak if they find any problem like this, they should inform their elders and trust worthy people around them and share their feelings about that event. Worksheets is given to children to describe their personal feelings about good events and bad events of their life. Another topic of bullying is also described to them with many story examples and also ask them to give their own examples which face during their school time or in any other location. It was proved very beneficial as most of the children participate and ask questions to clarify their ambiguity. During training, children also learn from lessons about what is bullying, what its effects, how to rescue oneself from being a victim of bullying. Their response show their level of understanding towards the topics of Programme. Few activities is also given to children by asking general questions from their life and also realize them to explain the problems with elders or with their trust worthy whom they believe. They are also guided to keep themselves safe and make others safe too; if they saw someone being bullied by any person, one should have to tell this to elder one and keep that person safe. The lesson about friendship is also delivered to them and realize them the importance of friendship in their life. It also contains activities in which children participate and also have some worksheets which describes their understanding regarding the topics.

**Session 5 stay safe programme lessons for children.** In this session, safe and unsafe events and situations are being discussed with children and suggesting them solutions what to do when

feel unsafe or unsecure. Rescue oneself from that problematic situation. In this session, lesson about different types of touch is also delivered to children. Researcher use different tools to describe every lesson gently; as touch is the sensitive and private topic so, doll is used to understand different types of touches and also the nature of touch in general. Which touch is bad and which touch is good, children also participate when asked them to list the touches that they feel disgust and make them uncomfortable and also list out some touches that are good and which they like. Children also share list of some touches that they called confuse touches; they should tell their elders about the nature of touch. Almost after every lesson, children learn the rule of stay safe for their life. The rue is to Say No, Get away and tell. Lesson also cover the nature of touch either the touch is appropriate or it is inappropriate. There is another lesson which is related to the nature of secrets and explain children about the nature of secrets. There are bad or good secrets, many daily life examples are given to children to understand and differentiate between the good bad the bad secret. Then, asked them to describe the nature of touch to elders if they feel them bad. If they have bad secrets they should tell their elders and say no to the bad secrets. Another lesson contains the major discussion related to strangers that what are strangers and how they misguide you or how to deal with a stranger when you are all alone. There are also some rules to deal with strangers that should be followed like, never take nay thing from strangers and never go with strangers, etc. the major purpose of lessons is to make children confident enough to speak up and tell elders or adults about the touch, bullying, secrets, etc. and never keep a touch a secret. Always tell others.

Session 6 stay safe programme lessons for teachers. Teachers also receive training from stay safe programme about their activeness in the classroom environment and they should listen every children carefully. If any child tell them any secret or any issue regarding their life, regarding touch, bullying, abuse, secrets, etc. or any other problems they should deal them carefully and if the matter is serious then they should contact with the higher authority or

counseling office or center so they would deal with the situation better. Teachers were also guided about the nature and types of abuse and how to handle every abuse appropriately like if a child is emotionally disturb, teacher should handle them appropriately by listen their issue carefully and use strategies to handle them. Teachers should also use this lessons again in the classroom in the spare time to make children confident to deal with issues carefully. Teachers also guide with many strategies that they must follow in the classroom environment. They should observe every child keenly to understand change in their behaviors.